CLINICAL TRIAL: NCT02707107
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Multiple Escalating Doses of Intravenous WCK 5222 (Zidebactam and Cefepime) in Healthy Adult Human Subjects
Brief Title: MED Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Intravenous WCK 5222 (Zidebactam and Cefepime) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wockhardt (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: W-5222-101
Record Dates: First submitted 2016-02-15; First posted 2016-03-14 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-08

CONDITIONS: Serious Gram-negative Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 3 g of zidebactam (1 g q8h) and 6 g of cefepime (2 g q8h) or 6 (Active Comparator): administered as IV infusions every q8h, over a period of 60 minutes.
  Interventions: Drug: Intravenous infusions of WCK 5222
- Placebo (Placebo Comparator): administered as IV infusions every q8h, over a period of 60 minutes.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Intravenous infusions of WCK 5222
  Arms: 3 g of zidebactam (1 g q8h) and 6 g of cefepime (2 g q8h) or 6
Drug: Placebo
  Arms: Placebo

SUMMARY:
Study to evaluate the safety, tolerability and pharmacokinetics of multiple escalating doses of intravenous WCK 5222 (Zidebactam and Cefepime) in healthy adult human subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Have a body mass index of 18 to 30 kg/m2 (both inclusive) calculated as weight (kg)/height(m2).
2. Resting supine blood pressure of 90 to 139 (systolic)/40 to 89 (diastolic) mmHg and a resting pulse rate of 40 to 100 beats per minute.
3. Calculated creatinine clearance ≥80 mL/min (Cockcroft-Gault method).
4. All values of hematology, serum chemistry, coagulation, and urinalysis showing no clinically significant deviations from normal as judged by the Principal Investigator.

Exclusion Criteria:

1. Participation in another investigational drug or device study or treated with an investigational product within 30 days or 5 half-lives, whichever is longer, before investigational product administration in this study.
2. History/evidence of clinically relevant pathology related to the cardiovascular system, central nervous system, respiratory tract, gastrointestinal tract, endocrinology, immunology, hematology or any other systemic disorder/major surgeries, that in the opinion of the Principal Investigator would confound the subject's participation and follow-up in the study.
3. History of clinically significant food or drug allergy, including known hypersensitivity to cefepime or any other related drugs.
4. History of Clostridium difficile induced diarrhea or infection within 1 year before screening.
5. Prior exposure to zidebactam.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-03; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment | 14 days

SECONDARY OUTCOMES:
Maximum plasma concentration | 7 days
Time to Cmax | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Quintiles, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No